CLINICAL TRIAL: NCT02801474
Title: Surgical Management of Posterior Malleolar Fractures Using the Direct or Indirect Reduction Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Jin XIONG, Director in the Department of Orthopaedics, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 115690
Record Dates: First submitted 2016-06-01; First posted 2016-06-15 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Posterior Malleolus Fractures
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- direct reduction (Experimental): Intervention: The posterior and lateral malleoli were accessed via a posterolateral approach with the patients in prone position. The fibular fracture was exposed and reduced anatomically in the first place. The posterior malleolus was then exposed between the fiexor halluces longus and peroneus longus interval. The posterior malleolar fragment was then reduced with reference to the typical metaphyseal-diaphyseal spike of the posterior malleolus. One-third tubular plate, reconstruction plate, or distal radius plate were applied spanning the fracture in a buttress mode. Cannulated screws could also be used.
  Interventions: Procedure: direct fracture reduction and fixation
- indirect reduction (Experimental): Intervention: After open reduction and internal fixation of lateral and medial malleolar fractures, the posterior malleolus was then reduced through ligamentotaxis with the ankle in dorsiflexion. One or two 4.0 mm cannulated screws were used to fix the posterior malleolar in anterior-to-posterior direction.
  Interventions: Procedure: indirect fracture reduction and fixation

INTERVENTIONS:
Procedure: direct fracture reduction and fixation — In the DR group, the posterior malleolar fracture was reduced and fixed in a direct way via a posterolateral approach with the patients in prone position.
  Arms: direct reduction
Procedure: indirect fracture reduction and fixation — In the IR group, the posterior malleolus was reduced through ligamentotaxis following open reduction and internal fixation of lateral and medial malleolar fractures. Percutaneous cannulated screws were used to fix the posterior malleolar in anterior-to-posterior direction.
  Arms: indirect reduction

SUMMARY:
Patients with a posterior malleolar fracture were recruited and assigned to the direct reduction (DR) group or the indirect reduction (IR) group. Following reduction and fixation of the fracture, the quality of fracture reduction was evaluated in radiograph and CT images. Functional outcome was evaluated at the last follow-up.

DETAILED DESCRIPTION:
Patients with a posterior malleolus fracture were recruited meeting the inclusion criteria of unstable and displaced posterior malleolar fractures requiring surgical management. Patients with open fractures or pathological fractures were excluded. Preoperative anteroposterior (AP), lateral, and mortise view radiographs as well as computed tomography (CT) scans were routinely obtained to evaluate the characteristic of the fracture. Patients were then assigned to the direct reduction (DR) group or the indirect reduction (IR) group. Following reduction and fixation of the fracture using the direct reduction technique or the indirect reduction technique, the quality of fracture reduction was evaluated in radiograph and CT images. Functional outcome,including AOFAS score, ankle range of motion were evaluated at the last follow-up.

ELIGIBILITY:
Inclusion Criteria:

* unstable ankle fracture requiring surgical intervention
* with posterior malleolar fracture

Exclusion Criteria:

* open fractures
* pathological fractures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2012-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
American Orthopaedic Foot and Ankle Society ankle-hindfoot score | 1 year

SECONDARY OUTCOMES:
ankle range of motion in degrees | 1 year
residual displacement of the posterior malleolus in mm | 3 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Jin XIONG, M.D., Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Nanjing Drum Tower Hospital, the Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shi HF, Xiong J, Chen YX, Wang JF, Qiu XS, Huang J, Gui XY, Wen SY, Wang YH. Comparison of the direct and indirect reduction techniques during the surgical management of posterior malleolar fractures. BMC Musculoskelet Disord. 2017 Mar 14;18(1):109. doi: 10.1186/s12891-017-1475-7. PMID 28292290